CLINICAL TRIAL: NCT07381478
Title: Effect of 3°C Saline Irrigation Toward the Duodenal Papilla to Prevent Post-ERCP Pancreatitis: Protocol for a Multicenter, Controlled, Randomized, Patient-Blinded Trial in Bogotá, Colombia.
Brief Title: 3°C Saline Injection at the Duodenal Papilla to Prevent Post-ERCP Pancreatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: Hospital San Rafael de Facatativá (Unknown)
Responsible Party: Principal Investigator, Juan Pablo Alzate, Clinical research institute investigator, Universidad Nacional de Colombia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Act 25 august 2025
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cold Saline Papillary Irrigation (3°C) (Experimental): At the end of ERCP, 250 mL of sterile saline at 3°C is instilled onto the duodenal papilla in five 50-mL aliquots through the endoscope working channel, with aspiration between aliquots to enhance the local effect.
  Interventions: Procedure: Topical Cold Sterile Saline Irrigation of the Duodenal Papilla (3°C)
- Standard ERCP (Usual Care) (Active Comparator): Standard ERCP performed with no additional saline instillation. Usual prophylaxis may be used when clinically indicated (e.g., rectal NSAIDs, lactated Ringer's hydration, prophylactic pancreatic stent in high-risk cases) and is recorded.
  Interventions: Other: Standard ERCP (Usual Care)

INTERVENTIONS:
Procedure: Topical Cold Sterile Saline Irrigation of the Duodenal Papilla (3°C) — 250 mL of 3°C sterile saline administered in five 50-mL aliquots directed to the papilla via the endoscope working channel at ERCP completion, with aspiration between aliquots; saline temperature is verified immediately before administration
  Arms: Cold Saline Papillary Irrigation (3°C)
Other: Standard ERCP (Usual Care) — Standard ERCP performed with no additional saline instillation. Usual prophylaxis may be used when clinically indicated (e.g., rectal NSAIDs, lactated Ringer's hydration, prophylactic pancreatic stent in high-risk cases) and is recorded.
  Arms: Standard ERCP (Usual Care)

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is an endoscopic procedure used to diagnose and treat problems in the bile ducts and pancreas. One of its most common complications is **post-ERCP pancreatitis**. This multicenter randomized clinical trial will evaluate whether **cooling the duodenal papilla** with **sterile saline at 3°C** immediately after ERCP can reduce the risk of post-ERCP pancreatitis compared with standard ERCP care.

Adults **≥18 years** with a **native papilla** scheduled for diagnostic or therapeutic ERCP at **three high-complexity university hospitals in Bogotá/Cundinamarca (Colombia)** will be randomized **1:1** to: (1) **intervention**-instillation of **250 mL** of **3°C sterile saline** in **five 50-mL aliquots** directed to the papilla through the endoscope working channel at the end of ERCP, with aspiration between aliquots; or (2) **control**-standard ERCP with no additional instillation. The saline temperature will be verified immediately before administration. Standard preventive measures (e.g., rectal NSAIDs, lactated Ringer's hydration, prophylactic pancreatic stent when clinically indicated) may be used per usual care and will be recorded.

The **primary outcome** is post-ERCP pancreatitis at **24 hours**, defined using Cotton criteria (new/worsening abdominal pain plus serum amylase or lipase ≥3× the upper limit of normal). Secondary outcomes include pancreatitis severity, other ERCP-related complications, and safety through day 7 (including a telephone follow-up). Participants will be screened and consented before sedation; randomization occurs at the end of the ERCP; clinical assessment and labs are performed at 24 hours; follow-up continues through day 7.

Safety monitoring will include systematic assessment for potential effects related to local cooling (e.g., chills, duodenal spasm, mucosal bleeding at the instillation site, or clinically relevant hypothermia) at 2 and 24 hours, with surveillance for serious adverse events through day 7.

ELIGIBILITY:
**Inclusion Criteria:**

* Adults **18 years of age or older**
* **Native (unmodified) duodenal papilla**
* Scheduled for **diagnostic or therapeutic ERCP**

**Exclusion Criteria:**

* **Inaccessible papilla** or papilla **surgically altered/modified**
* **Ongoing acute or chronic pancreatitis**
* **Pregnancy**
* **Ethical or medical contraindications to ERCP**
* **Lack of informed consent**

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-01-12 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Incidence of post-ERCP pancreatitis (PEP) at 24 hours | 24 hours after ERCP
  Proportion of participants with PEP defined by Cotton criteria: compatible abdominal pain plus serum amylase or lipase ≥3× upper limit of normal at 24 hours

SECONDARY OUTCOMES:
Incidence of moderate-to-severe post-ERCP pancreatitis | Up to Day 7 after ERCP
Abdominal pain assessment | 24 hours after ERCP

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital San Rafael de Facatativá, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Undecided